CLINICAL TRIAL: NCT06822361
Title: Assessment of Response to Vascular Filling by Uncalibrated Pulse Wave Contour Analysis in Beating Heart Cardiac Surgery
Brief Title: Uncalibrated Pulse Contour to Assess Fluid Responsiveness in Off Pump Cardiac Surgery
Acronym: UPC-OPCS
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/CHU/57; 2024-A02390-47 (Other: ID-RCB)
Record Dates: First submitted 2024-12-18; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: Coronary Surgery
Keywords: vascular filling; systolic ejection volume; uncalibrated pulse-wave contour analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to Compare the performance of uncalibrated pulse wave contour analysis compared with transesophageal echocardiography (TEE) to assess response to a vascular filling test during beating-heart coronary artery bypass surgery, in people over age of 18; hospitalized for scheduled beating heart bypass surgery The aim question is to evaluate the ability of a less invasive cardiac output monitor (uncalibrated pulse wave contour analysis) compared with a reference cardiac output measurement (transesophageal echocardiography) to enable optimization of vascular filling by good assessment of the response to vascular filling in a high-risk perioperative patient population.

As part of hemodynamic monitoring, every patient undergoing beating-heart coronary bypass surgery is fitted with a radial arterial catheter immediately after induction of anesthesia, enabling continuous measurement of blood pressure. Hemodynamic optimization in these patients also involves fitting a transesophageal ultrasound probe to optimize cardiac output using the various therapies available (vascular filling, vasopressors, inotropes).

A specific sensor (FloTrac°, Hemosphere, Edwards°) will be connected to the arterial pressure line to obtain a systolic ejection volume value by analyzing the contour of the uncalibrated pulse wave.

The hemodynamic management of the patient, and the decision to perform a vascular filling test, will be left to the discretion of the practitioner in charge of the patient in the operating room.

ELIGIBILITY:
Inclusion Criteria:

Patient :

* 18 years of age and older
* Hospitalized for scheduled beating-heart coronary bypass surgery
* Beneficiary of a social security plan
* Not opposed to participating

Exclusion Criteria:

* Patients undergoing surgery with extracorporeal circulation
* Patients with a history of surgery or intra-esophageal pathology contraindicating TEE
* Patient refusing to participate in the study
* Unavailability of TEE or uncalibrated pulse-wave contour device
* Minors
* Protected adults, adults unable to give consent and not under protective supervision
* Persons deprived of liberty, hospitalized without consent
* Pregnant women, parturients and nursing mothers
* Patients not affiliated to the social security system
* Emergency situations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient admitted to the cardiac surgery department for surgery under extracorporeal circulation
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Response to vascular filling | From enrollment to completion of chirurgy (24 hours)
  an increase of more than 10% (compared with basal value) in the sub-aortic VTI value measured in TEE after filling (gold standard).

IPD SHARING:
Plan to Share IPD: No